CLINICAL TRIAL: NCT02747264
Title: eRAPID Electronic Patient Self-Reporting of Adverse-events: Patient Information and aDvice: Feasibility Pilot Study in Radiotherapy
Brief Title: eRAPID Feasibility Pilot Study in Pelvic Radiotherapy
Acronym: eRAPID-RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Galina Velikova, Professor of Psycho-social and Medical Oncology/ Consultant in Medical Oncology, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RP-PG-0611-20008
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cancer
Keywords: eRAPID; PRO; PROM; Adverse event; QTool; CTCAE
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eRAPID intervention (Experimental): Participants in the intervention arm will receive training in using the eRAPID system to report their symptoms and side effects (at least on a weekly basis) from home via the internet whilst they are receiving treatment online and weekly for 6 weeks post treatment (a total of 12 weeks) and then at 18 & 24 weeks. Hospital staff will be able to review eRAPID reports and use the information during the consultation in clinic, when attending radiotherapy or answering phone calls. Alerts will also be sent to the relevant clinical team when severe symptoms are reported by patients.
  Interventions: Device: eRAPID
- Usual care (No Intervention): The Usual care patients act as a comparison to the patients using eRAPID. They complete a paper-based quality of life questionnaire at baseline and then 6, 12 and 24 weeks after. The researchers will also collect clinical process measures for this group including number of hospital contacts and admissions.

INTERVENTIONS:
Device: eRAPID — eRAPID is an online system for patients to self-report symptoms and AE during and after cancer treatments. eRAPID allows AE reporting from home or hospital and enables patient reported data to be integrated into existing EPR to allow for the reports to be used in routine care. In addition the system is capable of generating alerts for severe AE to the relevant clinical team and providing patient advice on managing mild and moderate AE.
  Arms: eRAPID intervention

SUMMARY:
The purpose of the Electronic Patient Self-Reporting of Adverse-events: Patient Information and aDvice (eRAPID) programme is to determine whether eRAPID (an online system for patients to self-report symptoms and side effects) can enhance patient care and improve the safe delivery of cancer treatments. The investigators hypothesise that patient symptoms will be detected earlier with more timely admissions and a reduction in overall hospital contacts. It is predicted that staff will save time recording symptoms and side effects and will be able to focus attention during clinical contacts on more severe side effects. eRAPID is a cost-effective approach to supporting patient self-management and reducing hospital/General Practitioner (GP)/community contacts.

The majority of the research will be run with systemic patients. This particular part of the research is a feasibility study in radiotherapy (RT) patients to test the platform in a different patient group.

DETAILED DESCRIPTION:
eRAPID is an online system for patients to self-report symptoms and side effects (known as adverse events or AE) during and after cancer treatments. eRAPID allows AE reporting from home or hospital and enables patient reported data to be integrated into existing Electronic Patient Records (EPR) to allow for the reports to be used in routine care. In addition the system is capable of generating alerts for severe AE to the relevant clinical team and providing patient advice on managing mild and moderate AE.

The investigators have developed the eRAPID system as a complex intervention by for use in patients undergoing pelvic RT specifically for prostate, cervical, vulval, anal, endometrial and rectal cancers. The investigators have done this by:

1. Integrating QTool questionnaire data with the Christie Manchester EPR; Clinical Web Portal (CWP) and in MOSAIQ (RT delivery system) in Leeds;
2. Developing tumour specific AE questionnaires and treatment algorithms for online reporting from home;
3. Mapping the current RT treatment pathways for these tumour groups via semi-structured interviews with staff and patients.

The overall aims of the eRAPID system are to improve the safe delivery of cancer treatments, enhance patient care and standardise documentation of AE within the clinical datasets.

AIMS AND OBJECTIVES In this feasibility pilot study, the investigators plan to test the complete eRAPID RT platform including patient and clinician interface. The investigators aim to examine feasibility, acceptability, and adherence to the intervention from the perspective of cancer patients and health professionals and explore the impact on patient care and quality of life. In addition, the investigators aim to determine effect sizes to inform the design and recruitment targets for a future randomised control trial.

STUDY SAMPLE AND RESEARCH DESIGN Adult patients attending St James' University Hospital Bexley Wing and the Christie Hospital Manchester starting radical treatment with RT for prostate cancer or chemo-RT for anal, rectal, cervical, endometrial and vulval cancer will be eligible to take part in this study.

This will be a prospective randomised parallel group design feasibility study with repeated measures and mixed methods. Participants will be randomised (following a 1:1 randomisation strategy) to receive the eRAPID intervention or usual care. The investigators aim to recruit a maximum of 168 patients to the study.

Participants in the intervention arm will receive training in using the eRAPID system to report their symptoms and side effects (at least on a weekly basis) from home via the internet whilst they are receiving treatment online and weekly for 6 weeks post treatment (a total of 12 weeks) and then at 18 & 24 weeks. Hospital staff will be able to review eRAPID reports and use the information during the consultation in clinic, when attending RT or answering phone calls. Alerts will also be sent to the relevant clinical team when severe symptoms are reported by patients. All patients will complete a paper-based quality of life questionnaire at baseline and then 6, 12 and 24 weeks after.

STUDY MEASURES

This study will use several outcomes to compare the eRAPID intervention with usual care:

Clinical outcomes and process of care measures For example the number of hospital contacts including admissions, clinic appointments, phone calls with hospital staff and changes to supportive medications and adjuvant chemotherapy dose change).

Patient-reported outcomes: Overall quality of life will be assessed using validated questionnaires and appropriate subscales (for example FACT-G 1 & EORTC-QLQ-C30 2 and Social function and symptoms scales and the EQ-5D 3).

Costs to patients and the NHS: Resource use will be assessed using patient questionnaires detailing contacts with GPs/community services, hospital visits and patient incurred costs, and others identified from use of resource forms.

Patient and staff interviews: Semi-structured staff, patients and carer interviews will be conducted to explore experiences of using the eRAPID intervention and any recommendations for improvement.

FINDINGS Overall findings will determine the value of the eRAPID intervention for supporting the care of patients receiving RT with or without concurrent chemotherapy as primary cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or over) attending St James' University Hospital or the Christie Hospital Manchester who have been:
* Diagnosed with prostate cancer requiring radical radiotherapy treatment (including radiotherapy +/- brachytherapy boost) Or
* Diagnosed with anal, rectal, cervical, endometrial or vulval cancer requiring chemo-radiotherapy.
* Able and willing to give informed consent
* Able to read and understand English
* Access to the internet at home or on a smart device

Exclusion Criteria:

* Patients taking part in other clinical trials involving the completion of extensive patient reported outcome or quality of life measures
* Patients exhibiting overt psychopathology/cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with self-reported outcome data at each time-point | 6 months
  Patients will complete a paper-based quality of life questionnaire
Proportion of missing data in patient outcome questionnaires | 6 months
  Patients will complete a paper-based quality of life questionnaire
Appropriateness of patient outcome questionnaires by assessing ceiling and floor effects ( quality of life questionnaire) | 6 months
  Descriptive statistics of returned questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Galina Velikova, Principal Investigator — The University of Leeds
Locations (2):
- United Kingdom (2):
  - The Christie Hospital, Manchester, Greater Manchester
  - St James University Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler L, Harley C, Holch P, Keding A, Bamforth L, Warrington L, et al. Towards Safer Delivery and Monitoring of Cancer Treatments. Electronic Patient Self-Reporting of Adverse-Events: Patient Information and a aDvice (eRAPID). Psycho-Oncology. 2012;21:15.
- [Background] Holmes M HP, Rodgers Z Dickinson S, Davison S, Routledge J, Henry A, Franks K, Gilbert A, Velikova G Patient and relative attitudes to the implemetation of eRAPID (Electronic patients self-Reporting of Adverse-events: patients Information and aDvice) during and after pelvic radiotherapy: a wualitative interview study. Psycho-oncology. 2016.
- [Background] Rogers Z HP, Homes M, Davidson S, Routledge J, Henry A, Franks K, Gilbert A, Dickinson S, & Velikova G. . Health care professional (HCP) attitudes to the implemntation of eRAPID (Electronic patient self-Reporting of Adverse-events: Patient Information and aDvice) during and after pelvic radiotherapy: a qualitative interview study. Psycho-oncology. 2016.
- [Background] Holch P, A, Henry, K, Franks , S, Davidson , A, Gilbert , J, Routledge , E, Ingleson, A, Albutt & G, Velikova Instruments to record acute and late adverse events (AE) associated with radical prostate cancer treatment for remote monitoring in clinical practice: A systematic review of randomised controlled trials (RCT). . Psycho-Oncology. 2015;24:1-15
- [Background] Holch P, Davidson S, Routledge J, Henry A, Franks K, Gilbert A, et al. OC-0416: eRAPID: Electronic self-report and management of adverse-events for radical prostate radiotherapy (RT) patients. Radiotherapy and Oncology. 2015;115, Supplement 1:S202.
- [Derived] Holch P, Absolom KL, Henry AM, Walker K, Gibson A, Hudson E, Rogers Z, Holmes M, Peacock R, Pini S, Gilbert A, Davidson S, Routledge J, Murphy A, Franks K, Hulme C, Hewison J, Morris C, McParland L, Brown J, Velikova G. Online Symptom Monitoring During Pelvic Radiation Therapy: Randomized Pilot Trial of the eRAPID Intervention. Int J Radiat Oncol Biol Phys. 2023 Mar 1;115(3):664-676. doi: 10.1016/j.ijrobp.2022.09.078. Epub 2022 Oct 12. PMID 36241128
- [Derived] Holch P, Pini S, Henry AM, Davidson S, Routledge J, Brown J, Absolom K, Gilbert A, Franks K, Hulme C, Morris C, Velikova G; eRAPID radiotherapy work group. eRAPID electronic patient self-Reporting of Adverse-events: Patient Information and aDvice: a pilot study protocol in pelvic radiotherapy. Pilot Feasibility Stud. 2018 Jun 5;4:110. doi: 10.1186/s40814-018-0304-6. eCollection 2018. PMID 29992040